CLINICAL TRIAL: NCT00224744
Title: Prospective and Randomized Study to Evaluate Interest of Ultracision Use in Inguinal Lymph Nodes Curage.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05 DIVE 03
Record Dates: First submitted 2005-09-22; First posted 2005-09-23 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2013-06

CONDITIONS: Vulvar Neoplasms; Skin Neoplasms
Keywords: Vulvar Neoplasms; Skin Neoplasms; Ultracision; Lymphadenectomy
MeSH Terms: conditions — Vulvar Neoplasms; Skin Neoplasms

ARMS (2):
- Classical surgical Inguinal curage (Active Comparator): Classical Inguinal curage
  Interventions: Device: classical lymphadenectomy
- Ultracision surgical Inguinal curage (Experimental)
  Interventions: Device: ultracision

INTERVENTIONS:
Device: ultracision — Surgery by Ultracision
  Arms: Ultracision surgical Inguinal curage
Device: classical lymphadenectomy — classical lymphadenectomy
  Arms: Classical surgical Inguinal curage

SUMMARY:
The purpose of this study is to evaluate the decrease of post-operative morbidity in inguinal lymphadenectomies realised for vulvar tumors and inferior limb skin tumors by use of Ultracision with regard to classical operative techniques.

ELIGIBILITY:
Inclusion Criteria:

* Vulvar neoplasm, inferior limb's skin malignant tumours, with an inguinal curage indication.
* Age ≥ 18 years
* Hematological functions : leucocytes > 1500/mm3, hemoglobin > 8 g/dl, blood platelets > 150000/mm3.
* Well informed written consent signed by the patient
* Negative pregnancy test for female patient of child-bearing potential.

Exclusion Criteria:

* Preliminary surgery of inguinal cavity (sentinel lymph node removal accepted)
* Massive lymph node invasion with femoro-vessels attack
* Inclusion in another study (excepted study turned to inguinal lymph node)
* Pregnant or nursing women
* Patient under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the decrease of post-operative morbidity. | 2012

SECONDARY OUTCOMES:
To study differences between the two techniques according to : operative duration ; operative difficulties ; quantity of drainage ; hospitalization's duration ; necessity of local care ; number of consultations ; medical and economical assessment. | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Denis Querleu, Pr, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - Institut Paoli-Calmettes, Marseille
  - Institut Claudius Regaud, Toulouse